CLINICAL TRIAL: NCT05775536
Title: Detection of Acetylsalicylic Acid and Omega-3 Fatty Acids in Schirmers' Test Strips Using Mass Spectrometry and Correlations With Tear Film and Blood Flow Parameters in Healthy Adults: an Open-label Pilot Study
Brief Title: Detection of Acetylsalicylic Acid and Omega-3 Fatty Acids in Schirmers' Test Strips Using Mass Spectrometry
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Doreen Schmidl, Assoc. Prof. Dr. Doreen Schmidl, PhD, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: OPHT-300920
Record Dates: First submitted 2023-02-24; First posted 2023-03-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aspirin® 500 mg tablets (Experimental): Dose: 1 tablet per day starting from visit 2 until visit 3, intake in the evening Ingredients: 500 mg acetylsalicylic acid, Cellulose powder, maize starche
  Interventions: Drug: Aspirin 500Mg Tab
- Dr. Böhm® Omega 3 complex 870 mg (Experimental): Dose: 2 tablets per day starting from visit 2 until visit 3, intake in the evening
  Interventions: Dietary Supplement: Dr. Böhm® Omega 3 complex 870 mg

INTERVENTIONS:
Drug: Aspirin 500Mg Tab — Dose: 1 tablet per day starting from visit 2 until visit 3, intake in the evening
  Arms: Aspirin® 500 mg tablets
Dietary Supplement: Dr. Böhm® Omega 3 complex 870 mg — Dose: 2 tablets per day starting from visit 2 until visit 3, intake in the evening
  Arms: Dr. Böhm® Omega 3 complex 870 mg

SUMMARY:
Evaluation of tear fluid production using Schirmers' tests is a well-known and frequently used examination method in ophthalmology. Schirmers' test objectively indicates the tear fluid production over five minutes by insertion of a filter paper strip in the lower conjunctival fornix. Commonly, this method is used to quantify tear fluid production, but not tear fluid composition. The development of novel, very precise analytical methods opens up new possibilities in the use and application of Schirmers' test strips. A recently introduced analytical method is mass spectrometry. This method allows the detection and quantification of proteins, lipids, and metabolites in very low amounts of samples. Whether systemically ingested agents such as omega-3 fatty acids or acetylsalicylic acid can be detected in tear fluid using this method remains unclear. The aim of this study is to investigate the detectability of 2 different agents (acetylsalicylic acid and omega-3 fatty acids) in Schirmers' test strips from healthy subjects after intake for 1 week by use of untargeted mass spectrometry. Participating healthy subjects will receive either acetylsalicylic acid or omega-3 fatty acids.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age of at least 18 years to 60 years
* Written informed consent prior to study-related procedures
* Normal ophthalmic findings
* No use of eye drops including topical lubricants in the 4 weeks before screening

Exclusion Criteria:

* Participation in a clinical trial in the 3 weeks preceding the study
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Presence or history of a severe medical condition as judged by the clinical investigator
* Intake of any drugs or dietary supplements within three weeks before the first study day (except contraceptives)
* TFBUT <10 sec.
* Glaucoma in the medical history
* Ocular infection or clinically significant inflammation
* Ocular surgery in the 3 months preceding the study
* Pregnancy, planned pregnancy or lactating
* Known hypersensitivity to any component of the study medication

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Concentration of omega-3 fatty acids/ASS detectable in Schirmer's tear strips using mass spectrometry | one week
Change of nAUC (normalised area under the curve) of tear fluid metabolics from baseline to follow-up visit using mass spectrometry | one week

SECONDARY OUTCOMES:
To evaluate the influence of omega-3 FA/ASS on lipid layer thickness | one week
  Lipid layer thickness will be measured by LipiView and expressed as nanometers
To evaluate the influence of omega-3 FA/ASS on corneal sensation | one week
  Corneal sensation as measured by a Cochet-Bonnet aesthesiometer will be expressed as milimeters
To evaluate the influence of omega-3 FA/ASS on tear film break up time | one week
  Tear film break up time will be measured clinically and expressed as seconds
To evaluate the influence of omega-3 FA/ASS on Schirmer-1 test | one week
  Schirmer-1 test will be expressed as milimetres/5 minutes
To evaluate the influence of omega-3 FA/ASS on choroidal perfusion | one week
  choroidal perfusion will be measured using a LSFG device and expressed as mean blur rate
To evaluate the influence of omega-3 FA/ASS on central macular thickness | one week
  central macular thickness will be measured by OCT and expressed as µm
To evaluate the influence of omega-3 FA/ASS on vessel density as assessed by optical coherence tomography angiography | one week
  vessel density will be measured by OCTA
To evaluate the influence of omega-3 FA/ASS on tear film osmolarity | one week
  tear film osmolarity will be measured by TearLab and expressed as mOsm/L
Concentration of omega-3 fatty acids/ASS detectable in finger sweat samples and blood samples using mass spectrometry | one week

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Department of Clinical Pharmacology, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided